CLINICAL TRIAL: NCT05875077
Title: The Effect of Propofol Versus Dexmedetomidine on the Incidence of Postoperative Nausea and Vomiting in Ureteroscopic Procedures Under Spinal Anesthesia
Brief Title: Propofol Versus Dexmedetomidine on the Incidence of Postoperative Nausea and Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Beshoy Atef Nagiub, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-62-2022
Record Dates: First submitted 2023-04-03; First posted 2023-05-25 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol group (Experimental): will receive propofol infusion.
  Interventions: Drug: Propofol
- Dexmedetomidine group (Experimental): will receive dexmedetomidine infusion.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — compare the effects of dexmedetomidine infusion to propofol infusion during spinal anesthesia, on the incidence of postoperative nausea and vomiting in patients undergoing ureteroscopic procedures under spinal anesthesia.
  Arms: Dexmedetomidine group
Drug: Propofol — compare the effects of dexmedetomidine infusion to propofol infusion during spinal anesthesia, on the incidence of postoperative nausea and vomiting in patients undergoing ureteroscopic procedures under spinal anesthesia.
  Arms: Propofol group

SUMMARY:
Post-operative nausea and vomiting are a leading cause of recovery room delays and low patient satisfaction. Complications such as suture line tension, wound hemorrhage and dehiscence, elevated intracranial pressure, pulmonary aspiration, dehydration, and electrolyte imbalance have been linked to nausea and vomiting.

Many studies were done to explore the effects of propofol and dexmedetomidine on the incidence of post operative nausea and vomiting (PONV). In this study, we will compare propofol infusion to dexmedetomidine infusion on the incidence of PONV in patients undergoing ureteroscopic procedures under spinal anesthesia in the age group from 18 to 60 years with more than one risk factor for PONV (female, history of PONV, non-smoking).

DETAILED DESCRIPTION:
In regional anesthesia, the mechanism of postoperative nausea and vomiting through the effect of hypotension is extremely common. Low blood pressure can cause ischemia in the brain stem, which activates the medulla's circulatory, respiratory, and vomiting centers. According to some researchers, hypotension causes gut ischemia and the release of emetogenic chemicals (such as serotonin) from the intestines. The function of the gastrointestinal tract is similarly altered by neuraxial anesthesia. Local anesthetics suppress the sympathetic nervous system, resulting in unopposed vagal action and gastrointestinal hyperactivity. The effectiveness of vagolytic drugs in relieving nausea during spinal anesthesia has been cited as proof of the mechanism's importance. During regional anesthesia, visceral discomfort is a powerful stimulator of emetic symptoms. Handling abdominal viscera stimulates sensory vagal fibers and activates the vomiting center, causing emesis.

Although the specific mechanism by which propofol operates as an antiemetic is unknown, a central mechanism for propofol's antiemetic activity appears to be the most likely, and a peripheral antiemetic effect has also been considered.

Because of its broad range of effects, which include anxiolytic, sedative, analgesic, anesthetic-sparing, sympatholytic, and hemodynamic-stabilizing qualities, dexmedetomidine is a powerful 2-adrenergic agonist with prospective applications in clinical anesthesia. The use of dexmedetomidine as an anesthetic adjuvant intraoperative has resulted in significant reductions in the use of opioids and inhalation anesthetics, as well as a decrease in the incidence of emergence agitation, a favorable recovery profile, and a decrease in postoperative pain without adverse hemodynamic effects.

The aim of this study is to compare the effects of dexmedetomidine infusion to propofol infusion during spinal anesthesia, on the incidence of postoperative nausea and vomiting in patients undergoing ureteroscopic procedures under spinal anesthesia.

Participants will be adults aged 18 to 60 years, scheduled for ureteroscopic procedures under spinal anesthesia.

Included participants will be patients aged 18 to 60 years with American Society of Anesthesiologists physical status (ASA) I-II scheduled for a ureteroscopic procedure with more than one risk factor for PONV (female, history of PONV, non-smoking) during our study time frame.

Excluded patients are those with contraindications to spinal anesthesia, including infection at the injection site, bleeding diathesis, known left ventricular outflow obstruction, hypovolemia, and increased intracranial pressure, history of allergy or hypersensitivity to propofol or dexmedetomidine, gastrointestinal diseases, e.g., gastroenteritis and gastric ulcers, ear diseases, e.g., infections of the middle and inner ear, liver cirrhosis, those who have received antiemetic drugs within 48 hours before surgery, those undergoing procedure taking more than two hours and patients unwilling to participate.

After being accepted into the study, participants' age, gender, weight, medications, special habits (e.g., smoking history), history of PONV, and any other comorbidity will be collected. All subjects will be fasting for 6-8 hours for solids and at least 2 hours for clear fluids. Routine monitoring devices (five lead electrocardiograms, non-invasive blood pressure, and pulse oximetry) will be installed when the patient arrives in the operating room, and baseline mean blood pressure, heart rate, and oxygen saturation data will be collected. Before spinal anesthesia, each patient will be given 500 mL of Ringer solution. In the sitting posture, a 25-gauge spinal needle is used to puncture the L3-L4 interspace under sterile conditions and via the midline route. After the cerebrospinal fluid (CSF) free flow, 12.5-17.5 mg of bupivacaine will be given intrathecally, and patients will be placed in a supine posture and remain horizontal for at least 10 minutes. Patients will be randomly assigned to one of three groups (propofol, dexmedetomidine, or control) and will begin receiving an infusion of either propofol (at a rate of 1 mg/kg/hour), dexmedetomidine (at a rate of 0.5 micrograms/kg/hour with no boluses), or nothing in the control group. Patients will be given 3 liters of oxygen per minute through a nasal cannula after spinal anesthesia. After the sensory block at the level of T10 is confirmed by the lack of sensitivity to pinprick, surgery will begin. The heart rate, oxygen saturation, pulse rate, and mean arterial blood pressure will all be recorded. Mean arterial blood pressure readings will be taken before and after the spinal every 10 minutes till the end of the procedure. Hypotension is defined as a drop in mean arterial blood pressure (more than 20% below baseline) following spinal injection, and it is treated by increasing intravenous fluid administration and administering 2.5-5 milligram increments of ephedrine I.V. (every 3-5 minutes) until the hypotension is resolved.

Intraoperatively and up to 6 hours after surgery, the frequency and severity of nausea and vomiting will be monitored using the PONV intensity scale. If the patient has had two or more bouts of nausea and vomiting, he will be given 10 mg of metoclopramide intravenously as a rescue antiemetic. Non steroidal anti inflammatory drugs (NSAIDS) will be used to provide analgesia post-surgery.

The Ramsay sedation scale (RSS) will be used to assess the patient's level of sedation, with the sedation score being recorded right before the study medicines are injected and then every 10 minutes until the patient is discharged from the recovery room. The RSS scores are assigned from 1 to 6, with 1 indicating anxious, agitated, and restless behavior, 2 indicating sedation-oriented and tranquil behavior, 3 indicating sedation response to commands, 4 indicating a brisk response to light glabellar tap, 5 indicating a sluggish response to light glabellar tap, and 6 indicating deep sedation with no response.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 60 years
* ASA physical status I-II
* Scheduled for ureteroscopic procedure
* With more than one Risk factor for PONV (female, history of PONV, non-smoking).

Exclusion Criteria:

* Patients with contraindications for spinal anesthesia including infection at the injection site, bleeding diathesis, known left ventricular outflow obstruction, hypovolemia, and increased intracranial pressure.
* History of allergy or hypersensitivity to propofol or dexmedetomidine.
* Gastrointestinal diseases e.g. gastroenteritis and gastric ulcers, ear diseases e.g. infections of middle and inner ear, liver cirrhosis.
* Those who have received antiemetic drugs within 48 hours before surgery.
* Operations lasting more than two hours.
* The patient's unwillingness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
primary outcome | 6 hours
  Number of PONV episodes in patients undergoing ureteroscopic procedures under spinal anesthesia

SECONDARY OUTCOMES:
secondry outcome | 2 hours
  heart rate
tertiary outcome | 2 hours
  arterial blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralaini Medical School, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456